CLINICAL TRIAL: NCT06114836
Title: Pathophysiological Evidence Driven Management of GERD in Neonatal ICU Infants: Randomized Controlled Trial
Brief Title: GERD Infant Feeding Therapeutics Trial (GIFT Trial)
Acronym: GIFT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Sudarshan Jadcherla, Principal Investigator, Innovative Feeding Disorders Research Program, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003300; 1R01DK136762-01 (NIH)
Record Dates: First submitted 2023-10-26; First posted 2023-11-02 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: GERD in Infants
Keywords: Proton Pump Inhibitor; pH Impedance; added rice formula
MeSH Terms: interventions — Omeprazole

STUDY DESIGN:
Intervention Model Description: Infants will be randomized to one of three arms: Natural maturation, Proton Pump Inhibitor (PPI) treatment, or Added rice (AR) formula. Subjects will be stratified and allocated 1:1:1 based on tube feeds (yes or no) and ARI (3-7% or >7%).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Natural maturation (No Intervention): Allows for time for infant maturation without treatment.
- Proton Pump Inhibitor (PPI) (Active Comparator): Omeprazole will be prescribed for 4 weeks using the dose of 1.5mg/kg/dose daily.
  Interventions: Drug: Omeprazole
- Added Rice (AR) Formula (Active Comparator): Added rice formula will be ordered as the infant diet for the 4-week treatment period.
  Interventions: Other: AR formula

INTERVENTIONS:
Drug: Omeprazole — Omeprazole will be the PPI prescribed for 4 weeks.
  Other Names: PPI
  Arms: Proton Pump Inhibitor (PPI)
Other: AR formula — Added rice formula will be ordered for 4 weeks.
  Arms: Added Rice (AR) Formula

SUMMARY:
The goal of this investigator-initiated, single-center, randomized controlled trial (RCT) is to compare the effects of four weeks of three therapies on clinical and mechanistic outcomes based on pH-Imp testing using a three-arm parallel design in NICU infants with objective GERD diagnosis. The three therapies being compared are natural maturation, proton pump inhibitor (PPI) use, and added rice (AR) formula use. The main goals are:

* to evaluate and compare the efficacy of the three commonly used treatment interventions used in the NICU for GERD in a randomized controlled manner with the primary endpoint of oral feeding success and absence of troublesome symptoms (as defined below).
* to characterize the mechanisms of primary end point (success or failure) using pH-Impedance metrics.

DETAILED DESCRIPTION:
In consented subjects, eligibility is determined after initial diagnostic 24-hour pH Impedance test. These subjects will be randomized to one of the 3 arms of the study (natural maturation, PPI, AR formula) for 4 weeks of treatment. A second 24-hour pH Impedance test will be done on therapy at 4 weeks or before discharge, whichever occurs first. Primary outcome will also be measured at 4 weeks or at discharge, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* NICU infants of any gestational age who are between 37 - 47 weeks postmenstrual age at inception of the study meeting the following requirements:

  * GERD diagnosis using pH-impedance criteria (Acid Reflux Index ≥ 3% plus at least one of the following: # GER events >70 / day, Symptom Associated Probability ≥ 95%, Discal Baseline Impedance < 900 Ω)
  * Full enteral feeds
  * No current GERD therapies

Exclusion Criteria:

* Known lethal chromosomal abnormalities or complex congenital syndromes
* Severe neurologic pathologies requiring neuroactive medications or neurosurgery
* Positive airway pressure or oxygen flow > 4 LPM
* Upper gastrointestinal malformations requiring surgery

Ages: 1 Day to 8 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 369 (Estimated)
Dates: Start 2024-03-14 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Achievement of primary outcome: Improvement or maintenance of oral feeding and/or absence of GERD symptoms (based on feeding method at inception) | At 4 weeks of therapy or discharge, whichever occurs first
  Achievement of the primary outcome will be measured by treatment group to determine efficacy. For subjects on full oral feeds at inception, the primary outcome will be met if there is maintenance of oral feeds AND absence of associated GERD symptoms. For subjects receiving any tube feeding at inception, the primary outcome will be met if there is improvement in oral feeding (ratio of oral to tube feeds) OR absence of troublesome symptoms. The metric for measuring the absence of troublesome symptoms will be vomiting <2 times/day or coughing <18 times/day.
Decrease in ARI on treatment | At time 2 study (4 weeks or prior to discharge, whichever is earliest)
  Change in acid reflux index from time one pH impedance study (prior to treatment) to time 2 pH impedance study (during treatment) will be compared among treatment groups.
Decreased frequency of GER events on treatment | At time 2 study (4 weeks or prior to discharge, whichever is earliest)
  Change in number of reflux events from time one pH impedance study (prior to treatment) to time 2 pH impedance study (during treatment) will be compared among treatment groups.
Improvement (Increase) in distal baseline impedance on treatment | At time 2 study (4 weeks or prior to discharge, whichever is earliest)
  Change in distal baseline impedance from time one pH impedance study (prior to treatment) to time 2 pH impedance study (during treatment) will be compared among treatment groups.
Decrease in symptom associated probability on treatment | At time 2 study (4 weeks or prior to discharge, whichever is earliest)
  Change in symptom associated probability from time one pH impedance study (prior to treatment) to time 2 pH impedance study (during treatment) will be compared among treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Sudarshan R sudarshan.jadcherla@nationwidechildrens.org, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospita, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Will revisit at a later date